CLINICAL TRIAL: NCT02221739
Title: Phase II Study of Combined Ionizing Radiation and Ipilimumab in Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of Combined Ionizing Radiation and Ipilimumab in Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00208
Record Dates: First submitted 2014-06-24; First posted 2014-08-20 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: lung cancer; NSCLC; lung; cancer; radiation; immunotherapy; metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Ipilimumab; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ipilimumab + radiotherapy (Experimental): Patients receive ipilimumab (Ipi) 3mg/kg i.v. over 90 minutes, within 24 hours of starting radiotherapy (RT) to the biopsied lesion, 6 Gy x5, later changed to 9.5 Gy x3 (conformally or by intensity modulated RT (IMRT) with image guidance to maximally spare normal tissue). Ipilimumab is repeated on days 22, 43 (for patients who consent to the first biopsy), and 64. Repeat biopsy is performed between day 22-29, and patients are re-imaged between day 81-88 and evaluated for response (defined as an objective response by irRC of the measurable metastatic sites outside the radiation field).
  Interventions: Drug: Ipilimumab; Radiation: Radiotherapy (IMRT or 3-D CRT)

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy
Radiation: Radiotherapy (IMRT or 3-D CRT)

SUMMARY:
The purpose of this study is to investigate how effective and how safe the combination of radiation therapy and an investigational medication targeting the immune system known as Ipilimumab in the treatment of metastatic non-small cell lung cancer (NSCLC).

The investigators would like to see if this combination of radiation and Ipilimumab can stimulate the body's immune system to stop the growth of tumors that are outside the field of radiation. The investigators would like see if using this combination of radiation therapy with Ipilimumab could help the body reject the patient's own tumor or at least help their immune system to maintain the disease stable and/or slow its growth.

Radiation therapy (RT) is currently a standard procedure for treatment of NSCLC. Ipilimumab is considered an investigational medication because it is not approved by the Food and Drug Administration (FDA) for the treatment of NSCLC. Ipilimumab has been approved by the FDA for the treatment of metastatic melanoma.

DETAILED DESCRIPTION:
Research Hypothesis:

1. Through a combination of local RT and ipilimumab an anti-tumor immune response is elicited at the irradiated site, as an in vivo, individualized immunization that is systemically effective, as reflected by objective responses outside the RT field (abscopal effect).
2. The immune response can be prospectively monitored among the treated patients.

Objective 1: Evaluate the safety and therapeutic efficacy of anti-cytotoxic T-lymphocyte-associated protein -4 mono clonal Antibody (anti-CTLA-4 mAb) and concurrent local RT in NSCLC patients with metastatic disease.

An open label phase II trial will evaluate the preliminary efficacy of the combination of Ipi and RT, applied to a single metastatic site. Efficacy is measured with respect to systemic tumor responses (abscopal response, outside the field of therapy) defined by immune-related Response Criteria (irRC) in all non-irradiated measurable lesions, as a demonstration of an effective anti-tumor immune response. Secondary endpoints include local response in the RT treated tumor, progression free survival, and overall survival.

Objective 2: Determine the effects of RT and anti-CTLA-4 mAb on development of anti-tumor immunity.

The investigators hypothesize that RT will convert the irradiated tumor into an in situ vaccine and elicit an endogenous tumor-specific cellular and humoral immune response, which in the presence of cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) blockade will promote immune-mediated destruction of the irradiated and abscopal metastases. Pre- and post-treatment tumor biopsies will be examined for changes in immune contexture, and blood for evidence of emerging anti-tumor immune responses. Associations with clinical response will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document;
2. Histologic diagnosis of metastatic NSCLC;
3. Any Kras or EGFR status is permitted;
4. Patients must have at least two distinct measurable metastatic sites, with one of at least 1 cm or larger in its largest diameter. Patients may have additional non-measurable metastatic lesions (e.g., bone metastases);
5. Patients must have prior treatment with at least one line of therapy for metastatic NSCLC. Any prior therapy is permitted except prior therapy with ipilimumab;
6. An interval of 2 weeks from last previous therapy is required;
7. Patients must have adequate organ and marrow function as defined by initial laboratory tests:

   * WBC ≥ 2000/uL
   * ANC ≥ 1000/uL
   * Platelets ≥ 50 x 103/uL
   * Hemoglobin ≥ 8 g/dL
   * Creatinine ≤ 3.0 x ULN
   * AST/ALT ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present.
   * Bilirubin ≤ 3.0 x ULN (except patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dL);
8. Performance status ECOG 0-1;
9. Men and women, ages > 18 years of age;
10. Life expectancy > 3 months;
11. Patients may have brain metastases if these are stable for at least 4 weeks, or greater than 2 weeks post gamma knife therapy and patients are not steroid dependent;
12. Brain Scan (CT/MRI) prior to enrollment
13. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of Ipi.

Exclusion Criteria:

1. Patients having no lesions outside the field of radiation thus nullifying the ability to measure an abscopal effect;
2. Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, progressive systemic sclerosis [scleroderma]), systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis];
3. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea;
4. Concomitant therapy with any of the following: Interleukin-2 (IL-2), interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids;
5. Prior therapy with ipilimumab or another anti-CTLA-4 antagonist;
6. Women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 8 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding;
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Chachoua, MD, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - NYU Clinical Cancer Center, New York, New York
  - NYU Langone Medical Center, Tisch Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab + Radiotherapy: Patients receive ipilimumab (Ipi) 3mg/kg i.v. over 90 minutes, within 24 hours of starting radiotherapy (RT) to the biopsied lesion, 6 Gy x5, later changed to 9.5 Gy x3 (conformally or by intensity modulated RT (IMRT) with image guidance to maximally spare normal tissue). Ipilimumab is repeated on days 22, 43 (for patients who consent to the first biopsy), and 64. Repeat biopsy is performed between day 22-29, and patients are re-imaged between day 81-88 and evaluated for response (defined as an objective response by irRC of the measurable metastatic sites outside the radiation field).
  Ipilimumab
  Radiotherapy (IMRT or 3-D CRT)
Period: Overall Study
Arm/Group | Ipilimumab + Radiotherapy
Started | 39
Completed | 21
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab + Radiotherapy
Number analyzed (Participants) | 39
Age, Customized [Median (Full Range); unit: years]
  Age | 68 [48 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 23
  Gender: Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 34
  Squamous Cell Carcinoma | 3
  Sarcomatoid | 1
  Neuroendocrine | 1

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy of Anti-CTLA-4 mAb and Concurrent Local RT in NSCLC Patients With Metastatic Disease.
Description: Tumor Response will be evaluated using the irRC best response (Partial Response (PR) + Complete Response (CR)). Modified WHO criteria will be used for measurement of tumors. The irradiated lesion will be excluded from the assessment of response.
Time Frame: 3 weeks - 6 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Radiotherapy
Number analyzed (Participants) | 21
Participants | 7

2. Secondary Outcome: Number pf Patients With Objective Radioactive Responses to Measure the Effects of RT and Anti-CTLA-4 mAb on Development of Anti-tumor Immunity Measured by T Cell Clone Frequency
Description: The study uses a comprehensive approach to analyze immunological changes that reflect both local and systemic responses, and investigate both general immune activation as well as tumor antigen-specific T- and B-cell responses. The activity of anti-CTLA-1 mAb is thought to be mainly dependent on modulating the quantity and quality of T-cells in cancer patients. A highly extensive analysis of the Cluster of differentiation 4 + (CD4+) and cluster of differentiation 8 + (CD8+) T-cell subsets will be characterized by multi-color flow Cytometry. To facilitate these analyses, serial blood samples will be collected for serum and peripheral blood mononuclear cells (PBMC) at different time points, where, a part of these samples will be used for DNA/RNA extraction. Optional tissue biopsies will be obtained from consenting patients.Tumor tissue will be tested for expression of seven antigens frequently expressed in NSCLC.
Time Frame: 3 weeks - 6 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Radiotherapy
Number analyzed (Participants) | 21
Participants
  Objective Radiographic Responses | 7
  Complete Responses (CR) | 2
  Partial Responses (PR) | 5

ADVERSE EVENTS:
Time Frame: 60 Months
Description: Adverse events as related to Ipilimumab or radiotherapy treatment. Grade of adverse event is shown: 1 - mild, 2 - moderate, 3 - Severe or medically significant but not immediately life-threatening, 4 - Life-threatening consequences, and 5 - Death related to AE.
Arm/Group | Ipilimumab + Radiotherapy
All-Cause Mortality (participants affected / at risk) | 17/39
Serious Adverse Events (participants affected / at risk) | 19/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab + Radiotherapy (N=39)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) — Patients that progressed or died before completion of treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab + Radiotherapy (N=39)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Alkaline Phosphotase (Hepatobiliary disorders) | 6 (6)
ALT (Hepatobiliary disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Anorexia (Psychiatric disorders) | 15 (15)
AST (Hepatobiliary disorders) | 5 (5)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cough (General disorders) | 3 (3)
Dehydration (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Dry Skin (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (Psychiatric disorders) | 9 (9)
Edema (Renal and urinary disorders) | 4 (4)
Fatigue (Psychiatric disorders) | 30 (30)
Fever (Psychiatric disorders) | 3 (3)
Hyperglycemia (Renal and urinary disorders) | 2 (2)
Hyperthyroid (Endocrine disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 4 (4)
Hypothyroid (Endocrine disorders) | 2 (2)
Hypoxia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Nausea (General disorders) | 5 (5)
Peripheral neuropathy (General disorders) | 3 (3)
Pruritis (General disorders) | 17 (17)
Rash (General disorders) | 13 (13)
Skin ulceration (General disorders) | 2 (2)
Tachycardia (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
50 dynamic changes of T cell clones in blood were the strongest response predictors, confirming 51 pre-clinical mechanistic data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT02221739/Prot_SAP_000.pdf